CLINICAL TRIAL: NCT02608281
Title: Clinical Study to Evaluate Diagnostic Accuracy of Low Dose Contrast Enhanced Dual Energy Mammography Imaging in Comparison to CE-MRI
Brief Title: Evaluation of Diagnostic Accuracy of Contrast Enhanced Dual Energy Mammography Imaging in Comparison to CE-MRI
Acronym: CEDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siemens Healthcare QT (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C00215154
Record Dates: First submitted 2015-10-09; First posted 2015-11-18 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer Diagnosis
Keywords: Spectral Mammography; Dual energy; Contrast enhanced
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CEDEM (Other): diagnostic contrast enhanced Dual Energy mammograms after Iodine based contrast media administration compared to CE MRI
  Interventions: Device: CONTRAST ENHANCED DUAL ENERGY (CEDEM)

INTERVENTIONS:
Device: CONTRAST ENHANCED DUAL ENERGY (CEDEM) — The CEDEM application requires the intravenous injection of iodide contrast agents. For each projection view (CC, MLO) a low and a high energy x-ray image will be acquired after Iodine based contrast medium administration. Patient will undergo CE MRI procedure.

SUMMARY:
Clinical study to evaluate diagnostic accuracy of low dose contrast enhanced dual energy mammography imaging (CEDEM+PRIME) in comparison with CE-MRI The primary objective of this clinical study is to assess diagnostic accuracy in breast cancer detection in Contrast Enhanced Dual Energy Mammography compared to CEMRI. Sensitivity and specificity will be compared for both modalities.

DETAILED DESCRIPTION:
STUDY OBJECTIVES The primary objective of this clinical study is to assess the value of low-dose CEDEM in comparison with CE-MRI. The diagnostic accuracy in breast cancer detection of low dose CEDEM will be evaluated.

Investigator plans to explore the diagnostic quality of 4 standard view bilateral dual energy subtracted images compared to CE-MRI in a blinded reader study. A goal is to evaluate, whether sensitivity and specificity of low-dose CEDEM are comparable with breast MRI.

Subjects will be asked before diagnostic workup to participate in this clinical study. Approximately 80 subjects scheduled for a diagnostic CE-MRI (i.e., based on screening mammography classified as BI-RADS® 0, 4 or 5), will be eligible to participate in this study and will undergo a follow up 4 view bilateral low dose contrast enhanced mammography procedure.

Radiologically, subjects included in the study population will have even distribution of masses, clusters of microcalcifications, and architectural distortions as given by the nature of breast cancer development.

The study population will include all breast compositions. Diagnostic CE-MRI Examination If eligible, subjects with a positive or incomplete screening mammogram (BI-RADS 0, 4 or 5) will undergo a CE-MRI of the breast. MRI examinations will be performed on a 3 Tesla scanner (Tim trio, Siemens) with a dedicated 16 channel breast coil. A combination of high temporal and high spatial resolution imaging protocol will be used. All patients will be examined in the prone position and contrast agent (0.2mmol / body weight, GD-DOTA) will be administered i.v. as a bolus followed by a 20 ml saline flush.

Both exams (CEDEM and CE-MRI) will be scheduled in the second week of the menstrual cycle in premenopausal women. Each suspicious lesion will undergo needle or surgical biopsy (after completion of the CEDEM+PRIME procedure). Imaging findings will be compared with findings of histology.

Diagnostic CEDEM+PRIME If eligible, subjects with a completed MRI procedure will undergo a 4 standard view (CC, MLO) bilateral CEDEM examination. Due to use of the grid-less PRIME acquisition technology the AGD is limited and lies in the range of a standard mammogram. The high energy images will be acquired with the titanium filter. All acquired images - including the unprocessed images - will be collected. Recombined CEDEM images will be created offline. Contrast agent is injected as a bolus of 2 ml/kg body weight of non-ionic iodine contrast media with a power injector at a rate of 3.5ml/s followed by a 25ml saline flush.

The CEDEM diagnostic procedure will be performed not later than 7 days and at least 24 hours after the CE-MRI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 21 years of age or older
* A screening mammogram classified as BI-RADS® 0, 4 or 5 followed by a diagnostic CE-MRI and a histological verification of a given lesions either by needle biopsy or open surgery
* Signed informed consent after receiving a verbal and written explanation of the purpose and nature of this clinical study

Exclusion Criteria:

* Pregnant or possible pregnant as well as lactating women
* Have mammographic evidence of previous breast surgery, prior radiation to the breast, needle projection or pre-biopsy markings are evident on the mammogram
* Breast implants
* Patients who will undergo neo-adjuvant chemotherapy (BI-RADS 6)
* Inmates or mentally disabled patient.
* Renal insufficiency or contrast agent allergy
* Patients who participated in other clinical studies within the last 12 months

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of contrast enhanced dual energy mammography for breast cancer diagnosis | 24 months
  Difference in accuracy of 11% comparing a 4-view contrast-enhanced dual energy imaging to CE-MRI assuming 11% discordant rate in the diagnosis

SECONDARY OUTCOMES:
sensitivity, specificity and the lesion-level ROC area. | 24 months
  The ROC area will be estimated from the BI-RADSS scores assigned by the readers to each suspicious lesion. The BI-RADS scores assigned by the readers in the interpretation of a CEDEM lesion will be used for the CEDEM+PRIME ROC area; the BI-RADS scores assigned by the readers in the interpretation of a CE-MRI case per lesion will be used for the CE-MRI ROC area. A receiver operating characteristic (ROC), or ROC curve, is a graphical plot that illustrates the performance of a binary classifier system as its discrimination threshold is varied. The curve is created by plotting the true positive rate (TPR) against the false positive rate (FPR) at various threshold settings

CONTACTS AND LOCATIONS:
Locations (1):
- Allgemeines Krankenhaus Wien, Vienna, Austria